CLINICAL TRIAL: NCT04878692
Title: Evaluation of a Cosmetic Product (Onco-Rash) to Preserve Skin Conditions When Using Anti-EGFR Cancer Therapies Which Are Known to Fragilize Epidermis
Brief Title: Evaluation of a Cosmetic Product to Preserve Skin Conditions When Using Anti-EGFR Cancer Therapies
Acronym: OPERA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 69HCL20_0519
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Head and Neck Neoplasms
Keywords: Skin Rash; anti-EGFR therapy; Cosmetic Product; Acne; Cancer patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Head and Neck Neoplasms; Exanthema; Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Onco-Rash arm (Experimental): In this arm label, patients will apply the Onco-Rash cream on selected zones (face, neck, thorax,…) twice a day, during 6 weeks.
  This arm will be compared to the Onco-Neutral arm, in which the Onco-Neutral cream will be applied on selected zones (face, neck, thorax,…) twice a day, during 6 weeks.
  Interventions: Drug: Application of Onco-Rash cream
- Onco-Neutre arm (Placebo Comparator): In this arm label, patients will apply the Onco-Neutre cream on selected zones (face, neck, thorax,…) twice a day, during 6 weeks.
  Onco-Neutral cream will be used as an experimental comparator to Onco-Rash cream.
  This arm will be compared to the Onco-Neutral arm, in which the Onco-Neutral cream will be applied on selected zones (face, neck, thorax,…) twice a day, during 6 weeks.
  Interventions: Drug: Application of Onco-Neutre cream

INTERVENTIONS:
Drug: Application of Onco-Rash cream — The cream "Onco-Rash" will be administered topically. The patient will be asked to apply the cream twice a day in the morning and evening for 6 weeks to clean, dry skin on selected target areas of the body, namely: the face, the front of the neck, the front of the chest, the back of the neck and the back of the chest. The product penetrates by gentle massage.
  Arms: Onco-Rash arm
Drug: Application of Onco-Neutre cream — The cream "Onco-Neutre" will be administered topically. The patient will be asked to apply the cream twice a day in the morning and evening for 6 weeks to clean, dry skin on selected target areas of the body, namely: the face, the front of the neck, the front of the chest, the back of the neck and the back of the chest. The product penetrates by gentle massage.
  Arms: Onco-Neutre arm

SUMMARY:
It is important for patients treated with anti-EGFR therapies to get access to cosmetic options to preserve their skin condition during treatment. Anti-EGFR therapies are known to fragilize epidermis and to provoke rashes; which often lead to treatment discontinuation.

The aim of this study is to demonstrate that the Onco-Rash cream is able to preserve skin condition without side effects. Decreasing skin toxicity is expected to improve patients' life and facilitate treatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Patient naive from anti-EGFR treatment (gefitinib, erlotinib, afatinib, cetuximab panitumumab, osimertinib, alectinib et crizotinib, etc).
* NSCLC (non-small cell lung cancer) patients eligible to anti-EGFR as first line treatment (gefitinib, erlotinib,afatinib, etc)
* Colorectal cancer patients eligible to anti-EGFR as first line treatment (cetuximab, panitumumab,….)
* Head and Neck/ENT (Ear, Nose Troat) cancer patients eligible to anti-EGFR as first line treatment (cetuximab,…)
* Signed informed consent
* Social security affiliation

Exclusion Criteria:

* Pregnant or Breastfeeding patient
* Patient in age to procreate without an efficient contraceptive method
* Patient with previous experience of allergic or irritative contact dermatitis to components of the studied product
* Patient with dermatologic conditions that cannot permit the study of skin toxicity of anti-EGFR
* Patients under radiotherapy 8 days prior the inclusion date
* Patient under immunotherapy 8 days prior the inclusion date
* Patient with local or systemic antibiotic treatment for acne 8 days prior the inclusion date
* Patient with antihistamines treatment 8 days prior the inclusion date
* Patients taking NSAIDs or corticoids as chronic medication or that took NSAIDs or corticoids 5 days prior the inclusion date
* Participation to another interventional study
* Patient with an altered ECOG (Eastern Cooperative Oncology Group) state ( >2)
* Patient deprived of liberty or subjected to guardianship
* Impossibility to track and follow patient for geographical, social or psychiatric reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the percentage of Onco-Rash failure by counting the number of patients with a rash grade ≥ 2 (NCI-CTCAE scale). | 6 weeks after the start of the anti-EGFR treatment.
  Measurement of Onco-Rash percentage of failure by counting the number of patients for whom a skin rash with a grade ≥ 2 (NCI-CTCAE scale) will occur between 0-6 weeks after the start of the anti-EGFR treatment. The introduction of an anti-inflammatory, a calming or an antibiotic treatment for acne will also be considered as failure.

SECONDARY OUTCOMES:
Timing of apparition of grade 1, 2 or ≥ 2 skin eruption: number of days between the start of the anti-EGFR treatment and the apparition of a skin eruption. | 6 weeks after the start of the anti-EGFR treatment.
  Comparison of timing of apparition of grade 1, 2 or ≥ 2 skin eruption between the Onco-Rash arm and the Onco-Neutral arm.
Percentage of patients with a grade 1, 2 or ≥ 2 skin eruption | 6 weeks after the start of the anti-EGFR treatment.
  Number of patients for whom a grade 1, 2 or ≥ 2 skin eruption have been reported
Percentage of patients for whom treatment for acne (anti-inflammatory or antibiotic) has been introduced | 6 weeks after the start of the anti-EGFR treatment.
  Number of patients for whom treatment for acne (anti-inflammatory or antibiotic) has been prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Julien PERON, MD, Principal Investigator — Institut de Cancérologie des Hospices Civils de Lyon - Service d'Oncologie médicale
Locations (1):
- Institut de Cancérologie des Hospices Civils de Lyon - Service Oncologie Médicale - Centre Hospitalier Lyon Sud, Pierre-Bénite, France